CLINICAL TRIAL: NCT00012337
Title: A Trial of ZD1839 (Iressa) in Patients With Advanced Renal Cell Carcinoma
Brief Title: ZD 1839 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068507; MSKCC-00125; NCI-1373
Record Dates: First submitted 2001-03-03; First posted 2004-03-17 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2002-03

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Some tumors need growth factors produced by the body's white blood cells to keep growing. Drugs such as ZD 1839 may interfere with the growth factors and cause tumor cells to die.

PURPOSE: Phase II trial to study the effectiveness of ZD 1839 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of ZD 1839 in patients with metastatic renal cell cancer. II. Determine the time to disease progression in patients treated with this drug. III. Determine the safety of this drug in these patients.

OUTLINE: Patients receive oral ZD 1839 once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 1 month.

PROJECTED ACCRUAL: A total of 16-46 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic renal cell carcinoma Bidimensionally measurable disease Bone metastasis as only site must have at least 1 bidimensionally measurable tissue mass by CT or MRI (e.g., expansile lesion) Radiologic evidence of disease progression or symptoms related to disease No brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL ALT/AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Other: No prior malignancy within the past 5 years unless potentially curatively treated or deemed at low risk for recurrence Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy and recovered No more than 1 prior biologic regimen No other concurrent biologic therapy Chemotherapy: At least 4 weeks since prior cytotoxic therapy and recovered No more than 1 prior cytotoxic regimen No concurrent cytotoxic therapy Endocrine therapy: At least 4 weeks since prior hormonal therapy and recovered No more than 1 prior hormonal regimen No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-01; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States